CLINICAL TRIAL: NCT05356390
Title: Comparative Effects of Stabilization Exercises and Muscle Energy Techniques on Pain and Disability in Sacroiliac Joint Patients
Brief Title: Comparative Effects of Stabilization Exercises and Muscle Energy Techniques in Sacroiliac Joint Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/Lhr/22/0107 Sana
Record Dates: First submitted 2022-04-28; First posted 2022-05-02 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Sacroiliac Joint Somatic Dysfunction
Keywords: pain; disability physical; muscle strength
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stabilization exercises (Experimental): Group A performed stabilization exercises for 4 weeks. In stabilization exercises, floor bridging, heel prop and alternate arm and leg exercises were administered in iliopsoas, gluteal and hamstring groups.
  Interventions: Other: Stabilization exercises
- Muscle energy techniques (Active Comparator): Muscle energy techniques were given to group B. These techniques are active form of manual therapy in which patient uses its own energy on request to aid in treatment.
  Interventions: Other: Muscle energy techniques

INTERVENTIONS:
Other: Stabilization exercises — Stabilization training is an active form of physical therapy designed to strengthen muscles to support the spine and help prevent lower back pain.
  Group A performed stabilization exercises for 4 weeks. In stabilization exercises, floor bridging, heel prop and alternate arm and leg exercises were administered in iliopsoas, gluteal and hamstring groups.
  On eligible participants baseline assessment was done,3 sessions were given 3days per week, post intervention assessment was taken at 4th week.
  Arms: Stabilization exercises
Other: Muscle energy techniques — Muscle Energy Technique (MET) is a is a form of manual therapy, widely used in Osteopathy, that uses a muscle's own energy in the form of gentle isometric contractions to relax the muscles via autogenic or reciprocal inhibition and lengthen the muscle.
  Muscle energy techniques were given to group B. These techniques are active form of manual therapy in which patient uses its own energy on request to aid in treatment.
  On eligible participants baseline assessment was done,3 sessions were given 3days per week, post intervention assessment was taken at 4th week.
  Arms: Muscle energy techniques

SUMMARY:
Sacroiliac joint is in pelvis. It links the iliac bone (pelvic) bone to the sacrum. This joint pain is due to hyper mobility or instability of the joint, it may also cause by damage to joint between the spine and hip. This pain is typically felt in the lower back, or hip and may radiate to groin area. The aim of this study will be to compare the effects of stabilization exercises and muscle energy techniques on pain and disability in patients with sacroiliac joint pain.

DETAILED DESCRIPTION:
A randomized clinical trial will be conducted at Ibn- e- Siena hospital and research institute Multan and in Bakhtawar Amin hospital Multan through convenience sampling technique on 30 patients which will be allocated through simple random sampling through sealed opaque enveloped into group A and group B. After giving common treatment of hot pack and transcutaneous electrical stimulation and assessing pre-treatment patient's condition Group A will be treated with stabilization exercises in which iliopsoas, gluteal and hamstring muscles will be stabilized. Total twelve sessions will be given as three sets three times per week for four weeks. Group B will be treated with muscle energy technique, this is active form of manual therapy in which patient will exert force against physiotherapist force through autogenic inhibition and reciprocal inhibition. (20% patient force against that applied by the physiotherapist and hold contractions for 10 seconds over 5 to 12 repetitions, 3 times per week for 4 weeks). Post-treatment assessment will be done after one month. Outcome measure will be conducted through pain and disability questionnaire after 6 weeks. Data will be analyzed using SPSS software version 21. After assessing normality of data by Shapiro -Wilk test, it will be decided either parametric or non-parametric test will be used within a group or between two groups. Stabilization exercises and muscle energy techniques will be applied for comparing their effectiveness in patients with sacroiliac joint pain.

ELIGIBILITY:
Inclusion Criteria:

* Both men and women age between 30-50 with positive Laslett's criteria. The Cluster of Laslett is a group of four test used for sacroiliac joint pain, the four tests are:

  1. Sacroiliac Distraction (Gapping) Test
  2. Thigh Thrust Test
  3. Sacroiliac Compression (Squish) Test
  4. Sacral Thrust test
* If a patient has three or more positive pain provocation tests, and then there is a 59% chance that the patient will have Sacroiliac joint pain.

Exclusion Criteria:

* Trochanteric bursitis
* Pelvic bone fracture
* Pelvic implants
* Pregnancy
* Lumbosacral disc herniation
* Sacroiliac joint inflammation
* Inflammatory bowel disease
* Malignancy

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2022-05-02 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-10-05 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | follow up at 4th week
  The Numeric Pain Rating Scale (NPRS) (an outcome measure) that is a unidimensional measure of pain intensity in adults, including those with chronic pain.
  The NPRS is a segmented numeric version in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of pain.
  The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").
  The NPRS takes <1 minute to complete The NPRS is a valid and reliable scale to measure pain intensity;
  * High test-retest reliability has been (r = 0.96 and 0.95, respectively)
  * For construct validity, the NPRS was shown to be highly correlated: correlations range from 0.86 to 0.95.
Modified Oswestry disability index | follow up at 4th week
  This questionnaire has been designed to give us information as to how your back or leg pain is affecting your ability to manage in everyday life. Please answer by checking ONE box in each section for the statement which best applies to you. A score of 0-20 reflects minimal disability, 21-40 moderate disability, 41-60 severe disability, 61-80 crippled, and 81-100 bed-bound.
  Each section is scored on a 0-5 scale, 5 representing the greatest disability. The index is calculated by dividing the summed score by the total possible score, which is then multiplied by 100 and expressed as a percentage. Thus, for every question not answered, the denominator is reduced by 5.

CONTACTS AND LOCATIONS:
Overall Officials: samrood Akram, MPhil, Principal Investigator — Riphah International University,Lahore
Locations (1):
- Bakhtawar Amin hospital Multan, Multan Khurd, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cho HJ, Kwak DS. Movement of the sacroiliac joint: Anatomy, systematic review, and biomechanical considerations. Proc Inst Mech Eng H. 2021 Mar;235(3):357-364. doi: 10.1177/0954411920978021. Epub 2020 Nov 30. PMID 33256545
- [Background] Sasaki T, Kurosawa D, Murakami E, Watanabe T. Physical therapeutic options for residual sacrotuberous ligament pain after treatment of sacroiliac joint dysfunction. J Phys Ther Sci. 2021 Sep;33(9):646-652. doi: 10.1589/jpts.33.646. Epub 2021 Sep 1. PMID 34539068
- [Background] Rashbaum RF, Ohnmeiss DD, Lindley EM, Kitchel SH, Patel VV. Sacroiliac Joint Pain and Its Treatment. Clin Spine Surg. 2016 Mar;29(2):42-8. doi: 10.1097/BSD.0000000000000359. PMID 26889985
- [Background] Barros G, McGrath L, Gelfenbeyn M. Sacroiliac Joint Dysfunction in Patients With Low Back Pain. Fed Pract. 2019 Aug;36(8):370-375. PMID 31456628
- [Background] Cohen SP, Chen Y, Neufeld NJ. Sacroiliac joint pain: a comprehensive review of epidemiology, diagnosis and treatment. Expert Rev Neurother. 2013 Jan;13(1):99-116. doi: 10.1586/ern.12.148. PMID 23253394
- [Background] Ahmed UA, Maharaj SS, Van Oosterwijck J. Effects of dynamic stabilization exercises and muscle energy technique on selected biopsychosocial outcomes for patients with chronic non-specific low back pain: a double-blind randomized controlled trial. Scand J Pain. 2021 Feb 24;21(3):495-511. doi: 10.1515/sjpain-2020-0133. Print 2021 Jul 27. PMID 33641272
- [Background] Sanika V, Prem V, Karvannan H. Comparison of Glutues Maximus Activation to Flexion Bias Exercises Along with MET Technique in Subjects with Anterior Rotated Sacroiliac Joint Dysfunction-a Randomised Controlled Trial. Int J Ther Massage Bodywork. 2021 Mar 1;14(1):30-38. eCollection 2021 Mar. PMID 33654504
- [Background] Garcia-Penalver UJ, Palop-Montoro MV, Manzano-Sanchez D. Effectiveness of the Muscle Energy Technique versus Osteopathic Manipulation in the Treatment of Sacroiliac Joint Dysfunction in Athletes. Int J Environ Res Public Health. 2020 Jun 22;17(12):4490. doi: 10.3390/ijerph17124490. PMID 32580480
- [Background] Sarkar M, Goyal M, Samuel AJ. Comparing the Effectiveness of the Muscle Energy Technique and Kinesiotaping in Mechanical Sacroiliac Joint Dysfunction: A Non-blinded, Two-Group, Pretest-Posttest Randomized Clinical Trial Protocol. Asian Spine J. 2021 Feb;15(1):54-63. doi: 10.31616/asj.2019.0300. Epub 2020 Jan 30. PMID 31992024
- [Background] Vaseghnia A, Shadmehr A, Attarbashi Moghadam B, Olyaei G, Hadian Rasanani DM-R, Khazaeipour Z. Effects of Muscle Energy Technique on Daily Activities and Lumbar Stiffness in Women With Sacroiliac Joint Dysfunction: A Randomized Controlled Clinical Trial Study. Journal of Modern Rehabilitation. 2019;13:23-30.